CLINICAL TRIAL: NCT02413294
Title: Sleep to Activate Mood Promotion- Intervention
Brief Title: Sleep to Activate Mood Promotion
Acronym: STAMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amanda Leggett, Postdoctoral Research Fellow, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HUM00094645
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Depression; Sleep Quality
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bright Light Intervention (Experimental): Before the bright light intervention is initiated (and during the intervention), participants will wear two wrist bands which measure sleep quality and activity levels- the Fitbit and actigraphy watches. These will be worn for two weeks to assess individuals' baseline levels of sleep quality and will continue to be worn during the intervention. Following the baseline period, the re-timer glasses will be introduced and worn for a period of 30 to 50 minutes a day for two weeks.
  Interventions: Device: Re-Timer glasses

INTERVENTIONS:
Device: Re-Timer glasses — Participants will wear the Re-timer glasses for 30 minutes a day according to their sleep chronotype in weeks 3 and 4 of the study.

SUMMARY:
The investigators are aiming to examine the acceptability and feasibility of a portable bright light therapy instrument to improve sleep disturbance in a preventive intervention for depression. The investigators will conduct an intervention that trials the use of bright light glasses called "re-timers" as a preventive intervention in older adults with sleep disturbance and subsyndromal symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older
* 6 or greater on the Pittsburgh Sleep Quality Index
* A score of 5 to 9 on the Patient Health Questionnaire-9 Depression Scale

Exclusion Criteria:

* Active suicidal ideation
* Presence of mania or bipolar disorder
* Presence of an eye disease
* Prescription of a photosensitizing medication
* Having previously had eye surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda N Leggett, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bright Light Intervention
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures are given for the study sample that completed study procedures.
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Asian American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11
Patient Health Questionnaire-9 [Mean (Standard Deviation); unit: units on a scale] — The PHQ-9 Depression Scale is a validated scale ranging from 0 to 27 with higher numbers representing greater severity of depressive symptoms, based on 9 questions with each question on a scale of 0 - 3.
  units on a scale
    Baseline | 5.6 (3.9)
    After 2 wks sleep tracking/prior to intervention | 3.7 (3.2)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index is a validated scale which measures self-reported sleep quality based on a wide variety of questions (duration, quality, disturbances, medication, etc.) and converts them to a scale which ranges from 0 to 21 where 6 or higher denotes poor sleep quality.
  units on a scale
    Baseline | 8.3 (4.1)
    After 2 wks sleep tracking/prior to intervention | 7.6 (3.7)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index measures insomnia severity on a scale from 0 to 28. A score of 15 or higher is indicative of clinical insomnia.
  Data for all 11 participants is provided at two baseline time points:
  prior to wearing a monitor at all, and after two weeks of wearing a monitoring device, prior to use of ReTimer glasses
  units on a scale
    Initial baseline measurement | 13.09 (4.85)
    After 2 wks sleep tracking/prior to intervention 3 | 11.86 (5.51)
Morningness/Eveningness Questionnaire [Count of Participants; unit: Participants]
  Morning type | 2
  Intermediate type | 8
  Evening type | 1

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index
Description: The Pittsburgh Sleep Quality Index is a validated scale which measures self-reported sleep quality based on a wide variety of questions (duration, quality, disturbances, medication, etc.) and converts them to a scale which ranges from 0 to 21 where 6 or higher denotes poor sleep quality.
Time Frame: two weeks after introduction of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
units on a scale | 7.0 (3.4)
Statistical Analysis 1: Comparison: Bright Light Intervention; The analysis, like the measures themselves, tracks the significance of the change from end of pre-intervention period to end of intervention period, so while only a single comparison group is listed, because it is all one population group, there are two sets of data for that group; Test type: Superiority; p = 0.37, Paired T test, 2-sided — This t-test analyzes the change in mean between the midpoint interview immediately prior to the start of the intervention and the follow-up interview at the conclusion of the intervention

2. Primary Outcome: Patient Health Questionnaire-9 Depression Scale
Description: The PHQ-9 Depression Scale is a validated scale ranging from 0 to 27 with higher numbers representing greater severity of depressive symptoms, based on 9 questions with each question on a scale of 0 - 3.
Time Frame: two weeks after introduction of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
units on a scale | 3.3 (2.3)
Statistical Analysis 1: Comparison: Bright Light Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.42, Paired T test, 2-sided

3. Primary Outcome: Insomnia Severity Index Sum Scores
Description: The Insomnia Severity Index measures insomnia severity on a scale from 0 to 28. A score of 15 or higher is indicative of clinical insomnia.
Time Frame: two weeks after introduction of intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
units on a scale | 11.36 (5.89)
Statistical Analysis 1: Comparison: Bright Light Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.65, Paired T test, 2-sided

4. Primary Outcome: Morningness-Eveningness Questionnaire
Description: The morningness- eveningness categories represent the time of day when a person is at their peak alertness.
Time Frame: two weeks after introduction of intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
Participants
  morning types | 3
  intermediate type | 8
  evening types | 0
Statistical Analysis 1: Comparison: Bright Light Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 1.0, Fisher Exact

5. Secondary Outcome: Actigraph Sleep Data: Minutes Asleep
Description: mean nightly sleep duration for each of the two-week periods: baseline and intervention
Time Frame: daily for 4 weeks- baseline and intervention period
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
minutes
  2 weeks monitoring prior to ReTimer use | 405.2 (27.9)
  2 weeks with ReTimer Glasses | 402.2 (24.5)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.65, Paired T test, 2-sided

6. Secondary Outcome: Actigraph: Number of Awakenings
Description: Actigraphy counts awakenings by using an accelerometer to assess motion during the night. The number of awakenings is the mean nightly number of awakenings during each of the two-week periods: baseline and intervention.
Time Frame: daily for 4 weeks- baseline and intervention period
Measure: Mean (Standard Deviation); unit: count of awakenings
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
count of awakenings
  2 weeks monitoring prior to ReTimer use | 22.1 (6.2)
  2 weeks with ReTimer Glasses | 22.4 (5.9)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.65, Paired T test, 2-sided

7. Secondary Outcome: Actigraph: Efficiency
Description: Sleep efficiency is calculated as a percentage reflecting the amount of time in bed spent asleep (time asleep/time in bed x 100). The mean for each of the two-week periods: baseline and intervention, is calculated.
Time Frame: daily for 4 weeks- baseline and intervention period
Measure: Mean (Standard Deviation); unit: percentage of time in bed spent asleep
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
percentage of time in bed spent asleep
  2 weeks monitoring prior to ReTimer use | 85.0 (4.5)
  2 weeks with ReTimer Glasses | 85.1 (4.0)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.94, Paired T test, 2-sided

8. Secondary Outcome: Fitbit Sleep Data: Sleep Duration
Description: mean nightly sleep duration in minutes for each of the two-week periods: baseline and intervention
Time Frame: daily for 4 weeks- baseline and intervention period
Measure: Mean (Standard Deviation); unit: Minutes asleep
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
Minutes asleep
  2 weeks monitoring prior to ReTimer use | 425.4 (33.6)
  2 weeks with ReTimer Glasses | 428.3 (36.6)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.81, Paired T test, 2-sided

9. Secondary Outcome: Fitbit Sleep Data: Night Awakenings
Description: mean nightly awakenings for each of the two week periods: baseline and intervention. Similar to the actigraph the Fitbit counts awakenings through an accelerometer which measures motion.
Time Frame: daily for 4 weeks- baseline and intervention period
Measure: Mean (Standard Deviation); unit: count of night awakenings
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
count of night awakenings
  2 weeks monitoring prior to ReTimer use | 13.4 (3.9)
  2 weeks with ReTimer Glasses | 15.8 (11.4)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.40, Paired T test, 2-sided

10. Secondary Outcome: Fitbit Sleep Data: Sleep Efficiency
Description: Sleep efficiency is calculated as a percentage reflecting the amount of time in bed spent asleep (time asleep/time in bed x 100).
Time Frame: daily for 4 weeks- baseline and intervention period
Measure: Mean (Standard Deviation); unit: percentage of time in bed spent asleep
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
percentage of time in bed spent asleep
  2 weeks monitoring prior to ReTimer use | 91.2 (2.2)
  2 weeks with ReTimer Glasses | 90.6 (4.1)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.46, Paired T test, 2-sided

11. Secondary Outcome: Self-Reported Sleep Diary: Time at Which Participants go to Bed
Description: Bed time represents the moment in time at which participants went to bed, measured on a revised clock where 6pm = 18, Midnight = 24 and 6am =30. Time between actual hours is calculated on a decimal basis, so an additional 6 minutes = .1. This revised clock is necessary in order to make means work properly in the nighttime hours. Otherwise, averaging between a 10pm bedtime and a 2am bedtime would give the impossible, inaccurate mean of being in the daytime between those two numbers.
Time Frame: daily for 4 weeks- baseline and intervention period to be compared
Measure: Mean (Standard Deviation); unit: hour (military time)
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
hour (military time)
  2 weeks monitoring prior to ReTimer use | 24 (1.4)
  2 weeks with ReTimer Glasses | 23.8 (1.3)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p < 0.01, Paired T test, 2-sided

12. Secondary Outcome: Self-Reported Sleep Diary: Time at Which Participants Wake up
Description: Wake time represents the moment in time at which participants awaken. Time between actual hours is calculated on a decimal basis so an additional 6 minutes = .1. so that 7.5 represents 7:30 a.m. and 7.8 represents 7:48 a.m.
Time Frame: daily for 4 weeks- baseline and intervention period to be compared
Measure: Mean (Standard Deviation); unit: hour (military time)
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
hour (military time)
  2 weeks monitoring prior to ReTimer us | 7.8 (1.8)
  2 weeks of ReTimer use | 7.5 (1.2)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.28, Paired T test, 2-sided

13. Secondary Outcome: Self-Reported Sleep Diary: Sleep Quality
Description: sleep quality is a participants' mean self-report for each of the two week periods: baseline and intervention. Sleep quality is reported for each night on a scale of 0 (very poor) to 4 (very good).
Time Frame: daily for 4 weeks- baseline and intervention period to be compared
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
units on a scale
  2 weeks monitoring prior to ReTimer use | 2.3 (0.5)
  2 weeks with ReTimer Glasses | 2.4 (0.6)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.67, Paired T test, 2-sided

14. Secondary Outcome: Self-Reported Sleep Diary: Night Awakenings
Description: mean number of night awakenings per person per night as reported in sleep diaries
Time Frame: daily for 4 weeks- baseline and intervention period to be compared
Measure: Mean (Standard Deviation); unit: Number of night awakenings
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
Number of night awakenings
  2 weeks monitoring prior to ReTimer use | 2.2 (1.3)
  2 weeks with ReTimer Glasses | 2.1 (1.0)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.56, Paired T test, 2-sided

15. Secondary Outcome: Self-Reported Sleep Diary: Sleep Duration
Description: nightly mean of length of sleep measured in minutes
Time Frame: daily for 4 weeks- baseline and intervention period to be compared
Measure: Mean (Standard Deviation); unit: Minutes asleep
Arm/Group | Bright Light Intervention
Number analyzed (Participants) | 11
Minutes asleep
  2 weeks monitoring prior to ReTimer use | 429.3 (28.2)
  2 weeks with ReTimer Glasses | 433.3 (56.5)
Statistical Analysis 1: Comparison: Bright Light Intervention; Pre-intervention period means are compared to intervention period means for all subjects; Test type: Superiority; p = 0.82, Paired T test, 2-sided

ADVERSE EVENTS:
Time Frame: Up to 29 days
Arm/Group | Bright Light Intervention
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes